CLINICAL TRIAL: NCT02726880
Title: Reducing Internet Gaming: A Pilot Psychotherapy Development Study
Brief Title: Reducing Internet Gaming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kristyn Zajac, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-114-3; P50DA009241 (NIH)
Record Dates: First submitted 2016-03-31; First posted 2016-04-04 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Behavior Therapy; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Referral for care (Active Comparator)
  Interventions: Behavioral: Referral for care
- Behavioral therapy (Experimental)
  Interventions: Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Behavioral therapy — 6-week behavioral intervention designed to assist with better monitoring and regulating the child's game playing behaviors.
  Arms: Behavioral therapy
Behavioral: Referral for care — Referral for mental health issues and family support services
  Arms: Referral for care

SUMMARY:
The fifth revision of the Diagnostic and Statistical Manual for Mental Disorders includes in its research appendix a potential new diagnosis-Internet gaming disorder. This condition primarily affects adolescent boys and young adult men, who rarely seek treatment on their own. More often, parents express concerns about their child's game playing behaviors. This psychotherapy development study will evaluate feasibility and effect sizes of an intervention designed to help parents reduce their child's gaming problems; the intervention allows for child participation, but it is geared toward parents, regardless of whether or not their child is willing to participate. A total of 40 parents concerned about their child's gaming behaviors will complete self and parental report inventories and structured diagnostic interviews regarding gaming, substance use and psychosocial functioning. Children who elect to participate will complete parallel versions of the instruments. Participants will be randomized to a control condition consisting of referral for mental health issues and family support services or to a 6-week behavioral intervention designed to assist with better monitoring and regulating the child's game playing behaviors. Gaming and other problems will be assessed pre-treatment, at the end of treatment and at a 4-month follow-up. This study will be the first to evaluate the reliability and validity of a parental version of the fifth revision of the Diagnostic and Statistical Manual for Mental Disorders criteria for internet gaming disorder in a clinical sample, and it will assess associations of internet gaming disorder with substance use, mental health conditions, and family functioning as well. This study will be the first randomized trial of an intervention designed to assist parents in reducing their child's gaming problems, and results will help guide future development of interventions for Internet gaming disorder. To evaluate the feasibility and acceptability of this intervention, the proportion of parents assigned to the intervention who complete 6 sessions will be examined, as will the proportion of youth who attend the sessions. Parent and child ratings of satisfaction with the intervention will be assessed. To examine the effect size of the intervention on reducing gaming, parental reports of proportion of days on which their child played games and durations of game playing will be compared between conditions, controlling for baseline indices.

ELIGIBILITY:
Inclusion Criteria:

* parent/guardian of a 10-22 year old residing in the same household >8 months/year
* reports significant problems with game playing

Exclusion Criteria:

* have a condition that may hinder study participation

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristyn Zajac, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Referral for Care | Behavioral Therapy
Started | 17 | 19
Completed | 14 | 16
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Referral for Care | Behavioral Therapy | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years is reported for the parents who participated in the study. The intervention was focused on child gaming behavior but the children were not required to participate in the study.
  years | 45.06 (9.28) | 50.58 (6.05) | 47.97 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 15 | 19 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 10 | 16 | 26
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 19 | 36
Number of days of gaming in the past week - reported by parent [Mean (Standard Deviation); unit: days] | 6.41 (1.73) | 6.42 (1.73) | 6.42 (1.46)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Complete All 6 Sessions
Description: Completion of sessions is an indicator of treatment acceptability and feasibility
Time Frame: 12 weeks
Population: This outcome is only reported for the Behavioral Therapy group because it is not relevant to the Referral to Care group. The Referral to Care group was not assigned to a structured 6 session intervention; thus, this outcome could not be measured in that group.
Measure: Number; unit: percentage of participants
Groups:
- Behavioral Therapy: 6 session behavioral therapy intervention designed to assist with better monitoring and regulating the child's game playing behaviors
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 19
percentage of participants | 78.9

2. Primary Outcome: Number of Days of Gaming in the Past Week - Reported by Parent
Description: Number of days of gaming is an indicator of the severity of the gaming problem.
Time Frame: 12 weeks
Population: The sample size for this analysis is smaller than the overall sample because several participants were lost to follow up.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Referral for Care | Behavioral Therapy
Number analyzed (Participants) | 14 | 18
days | 5.79 (2.19) | 5.06 (2.34)
Statistical Analysis 1: Comparison: Referral for Care vs Behavioral Therapy; Test type: Superiority; p = .296, ANCOVA; Number of days of gaming in the past week, measured at baseline, is included as a covariate in the model; F = 1.13

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Referral for Care | Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Referral for Care (N=17) | Behavioral Therapy (N=19)
hernia operation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Referral for Care (N=17) | Behavioral Therapy (N=19)
ER visit for car accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02726880/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02726880/ICF_001.pdf